CLINICAL TRIAL: NCT01187667
Title: Evaluation Study of a Delirium Prevention Policy Using Prophylactic Haloperidol in Critically Ill Patients With a High Risk for Delirium
Brief Title: Evaluation of Delirium Prevention in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Mark van den Boogaard, PhD, Radboud University Medical Center
Other Study IDs: 2010/May
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Delirium
Keywords: delirium; prevention; critical care; haloperidol
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Haloperidol prevention group: ICU patients with a high risk for delirium who are treated with haloperidol for preventive reason.
- Control group: Historical cohort group of patients (2008-2009)with a determined risk of 50% or more for delirium who were not treated with haloperidol for preventive reason.

SUMMARY:
Haloperidol is prescribed in high risk ICU patients concerning delirium (50% or more chance to develop delirium detected with the delirium prediction model PRE-DELIRIC, or patients with history of dementia or alcohol abuse)since the delirium protocol is changed and haloperidol is added as a prevention treatment we are gathering information what the effect is on several aspects of delirium

DETAILED DESCRIPTION:
Measurement the effect of haloperidol as delirium preventive intervention. Determining effect on:

- delirium incidence in the ICU - different subtypes of delirium - delirium free days in 28 days - days on the ventilator - length of stay on the ICU and In-Hospital - 28-day mortality - incidence of unexpected removal of tubes, and effect between different groups of patients. Safety of haloperidol concerning QT-time, extrapyramidal symptoms.

Data are compared with the data of a historical cohort

ELIGIBILITY:
Inclusion Criteria:

* Patients With Predicted Delirium Chance of >50% or history of dementia or alcohol abuse and treated with haloperidol

Exclusion Criteria:

* CAM-ICU is Not Applicable
* Patients Admitted 24hours or Shorter on the ICU, Patients Who Are Delirious Within 24 Hours After ICU Admission
* patients whereby haloperidol is contra-indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the ICU of a tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Delirium incidence | one year
  Delirium is diagnosed as minimal one positive CAM-ICU screening during complete ICU admission. Incidence rate is compared with historical cohort data

SECONDARY OUTCOMES:
duration of delirium days on mechanical ventilator Length of stay in the ICU and in-hospital in-hospital mortality incidence of unplanned removal of tube incidence of delirium subtypes | one year
  measured prospectively and determined in a CRF and compared with historical cohort data
Effect haloperidol on biomarkers | one year
  Biomarkers are measured in patients with high risk for delirium which are preventively treated with haloperidol

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] van den Boogaard M, Schoonhoven L, van Achterberg T, van der Hoeven JG, Pickkers P. Haloperidol prophylaxis in critically ill patients with a high risk for delirium. Crit Care. 2013 Jan 17;17(1):R9. doi: 10.1186/cc11933. PMID 23327295